CLINICAL TRIAL: NCT04940546
Title: Prospective Safety Study of Sintilimab Combined with XELOX Plus Bevacizumab for Preoperative Neoadjuvant Therapy of CRLM Patients with PMMR/MSS Status
Brief Title: Neoadjuvant Safety of Sintilimab + XELOX + Bevacizumab in PMMR/MSS CRLM Patients
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Yuhong Li, Clinical Professor, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: neoSXB-MSS-CRLM
Record Dates: First submitted 2021-06-18; First posted 2021-06-25 (Actual); Last update posted 2024-12-03 (Actual); Status verified 2024-11

CONDITIONS: Colorectal Cancer Metastatic
Keywords: Colorectal liver metastasis; pMMR/MSS; Sintilimab; XELOX; Bevacizumab
MeSH Terms: interventions — sintilimab; Oxaliplatin; Capecitabine; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Sintilimab + XELOX + Bevacizumab (Experimental): Patients receive Sintilimab + XELOX regimen every 3 weeks for 4 cycles and Bevacizumab every 3 weeks for 2 cycles.
  Details are as follows:
  Sintilimab: 200mg intravenously, d1 Oxaliplatin: 135mg/m2 intravenously, d1 Capecitabine: 2g/m2 orally, d1-14 for Bevacizumab: 7.5mg/kg intravenously, d1
  After neoadjuvant treatment, if there are no new lesions upon radiological and Multidisciplinary Team (MDT) assessment, radical surgery is performed within 6 weeks. If there are new lesions the surgical team will assess the optimal time for surgery.
  After surgery 4 cycles of XELOX regimen is advised for adjuvant therapy.
  Interventions: Drug: Sintilimab; Drug: Oxaliplatin; Drug: Capecitabine; Drug: Bevacizumab

INTERVENTIONS:
Drug: Sintilimab — Mode of administration: Intravenously
  Other Names: Anti-PD-1 monoclonal antibody IBI308
Drug: Oxaliplatin — Mode of administration: Intravenously
  Other Names: Eloxatin
Drug: Capecitabine — Mode of administration: Orally
  Other Names: Xeloda
Drug: Bevacizumab — Mode of administration: Intravenously
  Other Names: Avastin

SUMMARY:
This prospective, single arm study aims to evaluate the preoperative neoadjuvant safety of Sintilimab combined with XELOX plus bevacizumab in colorectal patients with liver metastasis and pMMR/MSS status.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

This preliminary prospective study aims to evaluate the safety of neoadjuvant treatment combination of Sintilimab, XELOX and bevacizumab and also asses safety during surgery of colorectal patients with liver metastasis and pMMR/MSS status.

SECONDARY OBJECTIVES:

To evaluate Pathological Remission Rate (pCR/MPR/PR rate), Objective Response Rate (ORR), Recurrence Free Survival (RFS) and Overall Survival (OS).

EXPLORATORY OBJECTIVES:

Analysis of liver metastasis before and after treatment to compare molecular and immunophenotypic changes.

OUTLINE:

Patients receive Sintilimab + XELOX regimen every 3 weeks for 4 cycles and Bevacizumab every 3 weeks for 2 cycles. After which if there are no new lesions upon assessment, radical surgery is performed within 6 weeks after neoadjuvant treatment. After surgery 4 cycles of XELOX regimen is advised for adjuvant therapy.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years old and ≤75 years old
* Histologically confirmed colorectal adenocarcinoma
* Radiologically and/or pathologically confirmed liver metastasis
* Immunohistochemistry and/or genetic testing confirmed pMMR/MSS
* Absence of extrahepatic metastasis confirmed by CT, MRI or PET/CT (if necessary)
* Primary lesion has been or can be removed by radical surgery
* Liver metastases can be resected (or using intraoperative radiofrequency) and is expected to achieve tumor-free status (NED) after surgery. Resectable liver metastases are defined explicitly as ① less than 5 metastatic lesions; ② R0 resection is achievable by resection or intraoperative radiofrequency; ③ Remaining liver volume is expected to be sufficient after surgery; ④ The following can be retained after resection: One hepatic vein, preserve blood flow in and out of the remaining liver, the bile duct, and at least 2 adjacent livers segments ⑤ There is no extrahepatic metastasis.
* Apart from surgical resection of the primary lesion, he/she has not received any anti-tumor treatment for liver metastasis (including chemotherapy, targeted drugs, interventional therapy, immunotherapy, radiotherapy, etc.)
* Normal hematological function (platelets>90×109/L; white blood cells>3×109/L; neutrophils>1.5×109/L)
* Serum bilirubin ≤ 1.5 times the upper limit of normal (ULN), transaminase ≤ 5 times ULN, alkaline phosphatase ≤2.5 ULN, No ascites, normal coagulation function, albumin ≥35g/L
* Child-Pugh classification of the liver is A
* Serum creatinine is less than the upper limit of normal (ULN), or the calculated creatinine clearance rate is greater than 50ml/min (using Cockcroft-Gault formula)
* ECOG score 0-1
* Life expectancy> 3 months
* Signed and written informed consent
* Willing and able to follow up until death or the end of the study or the study is terminated

Exclusion Criteria:

* Presence of distant metastases outside the liver after the diagnosis of colorectal cancer
* Liver metastases have been treated with chemotherapy, targeted drugs, intervention, immunotherapy, radiotherapy, etc.
* No surgical resection plan for liver metastases
* Received oxaliplatin-containing adjuvant chemotherapy in the past 1 year
* Any residual toxicity from previous chemotherapy (except for hair loss), such as peripheral neuropathy ≥NCI CTC v3.0 Grade 2
* Use of immunosuppressive drugs within 1 week before treatment, not including nasal sprays, inhalation or other local treatments, partial glucocorticoids or physiological doses of systemic glucocorticoids (i.e. not more than 10 mg/day prednisone or equivalent doses of other glucocorticoids) or use of corticoids to prevent contrast agent allergy
* Suffering from interstitial lung disease that requires steroid therapy
* Medical history of active autoimmune disease that needs symptomatic treatment within the past 2 years. Vitiligo, psoriasis, hair loss, or Grave's disease that do not require systemic treatment within the past 2 years, or hypothyroidism patients that only need thyroid hormone replacement therapy and type I diabetic patients requiring only insulin replacement therapy can be enrolled
* History of primary immunodeficiency
* Active tuberculosis
* Known history of allergies related to organ transplantation or hematopoietic stem cell transplantation
* Allergic to any monoclonal antibody or chemotherapeutic drug (fluorouracil, oxaliplatin) and its ingredients
* Have bleeding tendency or coagulopathy
* Patients with apparent symptoms of intestinal obstruction
* Hypertensive crisis or hypertensive encephalopathy
* Serious uncontrollable systemic complications such as infection or diabetes
* Clinically severe cardiovascular diseases such as cerebrovascular accident (within 6 months before enrollment), myocardial infarction (enrollment within the first 6 months), uncontrollable hypertension, unstable angina pectoris, heart failure (NYHA 2-4), arrhythmia requiring medical treatment
* Presence of central nervous system disease ( such as primary brain tumor, history of uncontrollable epilepsy, any brain metastases or stroke)
* Suffered from other malignant tumors in the past 5 years (except resected skin basal cell carcinoma and/or cervical carcinoma in situ)
* Received any drug treatment used for this study in the last 28 days
* Women who are pregnant and breastfeeding. Women of childbearing age who do not use or refuse to use effective non-hormonal contraceptive methods (intrauterine contraceptive ring, barrier contraception combined with spermicidal gel or female sterilization ) (<2 years after the last menstruation) or men with childbearing potential who are unable or unwilling to comply with the research protocol

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2021-06-16 (Actual); Primary Completion 2023-10-30 (Actual); Study Completion 2025-10-30 (Estimated)

PRIMARY OUTCOMES:
Adverse events | up to 24 months
  Number of patients with adverse events and severity according to NCICTCAE v5.0 during treatment period and using Clavien-Dindo classification of surgical complications for surgery.

SECONDARY OUTCOMES:
Pathological Remission Rate | up to 24 months
  Assessment of the absence of residual tumor pathologically
Objective Response Rate | up to 24 months
  Evaluation of changes in tumor size using the RECIST 1.1 criteria
Recurrence Free Survival | up to 24 months
  The length of time during and after the treatment of the disease, that a patient lives with the disease without recurrence
Overall Survival | up to 24 months
  The length of time from the start of treatment that patients diagnosed are still alive

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided